CLINICAL TRIAL: NCT07318753
Title: Shenzhen Hospital of Southern Medical University
Brief Title: A Clinical Study on The Use of DL-endopeptidase-producing Probiotics as an Adjunctive Therapy for Inflammatory Bowel Disease.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, Shenzhen Hospital of Southern Medical University, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShenzhenHZHW
Record Dates: First submitted 2025-11-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: gut microbiota; IBD; Crohn's disease; Ulcerative Colitis; DL-endopeptidase
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Take 2 grams of probiotic powder(LR607) daily from day 1 to day 5, and 4 grams daily from day 6 to day 90.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus CALM 607（LR607）
- Control (No Intervention): Take 2 grams of placebo daily from days 1 to 5, and 4 grams daily from days 6 to 90.

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus CALM 607（LR607） — Take 2 grams of probiotic powder(LR607) daily from day 1 to day 5, and 4 grams daily from day 6 to day 90.
  Arms: Experimental group

SUMMARY:
Through a series of studies,the investigators has discovered for the first time that gut microbiota-derived DL-endopeptidase is a core regulator of the NOD2 pathway. This research also reveals a novel etiological mechanism in which deficiency of gut bacterial DL-endopeptidase leads to dysfunctional NOD2 signaling, thereby promoting the pathogenesis of inflammatory bowel disease (IBD).( The findings have been published in Cell Host & Microbe and Nature Communications.) Based on this, the investigators has successfully screened a high DL-endopeptidase-producing active strain, Lactobacillus rhamnosus CALM 607 (abbreviated as LR607), from the traditional probiotic Lactobacillus rhamnosus.(Its unique advantages include: 1) Independent intellectual property rights (patent applied for);2) DL-endopeptidase production and NOD2 regulatory ability 2.7 times higher than that of the conventional strain LGG;3) Preclinical experiments have demonstrated its potential to alleviate intestinal inflammation.) The investigators' Phase I clinical trial (data pending publication) has confirmed that LR607 has good safety and tolerability in healthy volunteers, providing a safety foundation for subsequent clinical studies.

Therefore, the investigators aim to investigate the DL-endopeptidase-producing probiotic LR607 through randomized controlled clinical intervention studies, to evaluate its adverse effects in adjunctive therapy and comprehensively assess its impact on the gut microbiome-NOD2 pathway, intestinal inflammation, and the progression of IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ulcerative colitis (UC) Patients diagnosed with UC according to the 'Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (2023, Xi'an)'.

1. Patients with non-infectious UC initially diagnosed through laboratory tests, endoscopy, and pathological biopsy;
2. According to the latest guideline standards, clinically diagnosed with mild to moderate disease; defined as a modified Mayo score of 3-9 points; and classified as mild to moderate based on the modified Truelove and Witts severity classification;
3. In the active phase, with a clinical treatment plan using only mesalazine;
4. Voluntarily participating in this clinical trial, understanding, and signing the informed consent form.

2. Patients with Crohn's disease (CD) Patients diagnosed with Crohn's disease (CD) according to the 'Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (2023, Guangzhou)'.

1. Patients with non-infectious Crohn's disease (CD) initially diagnosed through laboratory tests, endoscopic examination, and pathological biopsy;
2. Clinically diagnosed as having mild to moderate disease according to the latest guideline standards, defined as a Crohn's Disease Activity Index (BestCDAI) score of 150-450;
3. Voluntarily participating in this clinical trial, having understood and signed the informed consent form.

Exclusion Criteria:

1. Patients with ulcerative colitis (UC) Patients diagnosed with UC according to the 'Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (2023, Xi'an)'.

1. Patients who have changed medication dosage or type in the past 2 months;
2. Patients who have the history of antibiotics, probiotics, or other medications affecting gut microbiota for non-target diseases within the past 2 months;
3. Patients who have the history of immunosuppressive drugs such as methotrexate or glucocorticoids ;
4. Patients who have the history of malignant tumors, other immune system diseases, or other serious chronic diseases;
5. Patients who have Concurrent active infections, including but not limited to obvious gastrointestinal bleeding, local or systemic infectious symptoms due to severe gastrointestinal ulceration or bleeding;
6. Pregnant or preparing for pregnancy and breastfeeding women;
7. Other situations deemed necessary to exclude by the researcher, for example: Simultaneous participation in other clinical interventional studies that may interact with this study.

2. Patients with Crohn's disease (CD) Patients diagnosed with Crohn's disease (CD) according to the 'Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (2023, Guangzhou)'.

1. Patients who have changed medication dosage or type in the past 2 months;
2. Patients who have the history of antibiotics, probiotics, or other medications affecting gut microbiota for non-target diseases within the past 2 months;
3. Patients who have the history of malignant tumors, other immune system diseases, or other serious chronic diseases;
4. Patients who have Concurrent active infections, including but not limited to obvious gastrointestinal bleeding, local or systemic infectious symptoms due to severe gastrointestinal ulceration or bleeding;
5. Pregnant or preparing for pregnancy and breastfeeding women;
6. Other situations deemed necessary to exclude by the researcher, for example: Simultaneous participation in other clinical interventional studies that may interact with this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Modified Mayo endoscopic score | 3 months
  Modified Mayo endoscopic score is divided into diarrhea, blood in stool, mucosal appearance, and physician assessment, each with a score of 0 to 3.
  * Clinical remission: score <2 with no individual subscore >1 ;
  * Mild activity: 3-5 points;
  * Moderate activity: 6-10 points;
  * Severe activity: 11-12 points

SECONDARY OUTCOMES:
The changes in gut microbiota structure | 3 months
  The gut microbiota composition was assessed through metagenomics before and after one and three months of taking probiotics or placebo. Compare and analyze the differences in gut microbiota structure at the three time points.
The Levels of NOD2 in the gut | 3 months
Endoscopic scoring（SES⁃CD/UCEIS） | 3 months
  SES⁃CD（4 parts: Including ulcer size, the proportion of intestinal segments with ulcers, the proportion of intestinal segments with non-ulcerative lesions, and strictures, each with a score of 0 to 3. Score the five intestinal segments (rectum, descending colon, transverse colon, ascending colon, and ileum) separately and calculate the total.）：
  * Remission phase: 0-2 points;
  * Mild activity: 3-6 points;
  * Moderate activity: 7-15 points;
  * Severe activity: ≥16 points; UCEIS（3 parts: Including vascular patterns(0-2 points), bleeding(0-3 points), and erosive ulcers(0-3points)）：
  * Remission phase: 0 points;
  * Mild activity: 1-3 points;
  * Moderate activity: 4-6 points;
  * Severe activity: 7-8 points;

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No